CLINICAL TRIAL: NCT01166997
Title: Randomized, Controlled Study Comparing EKOS EkoSonic Ultrasound Accelerated Thrombolysis to Anticoagulation in the Treatment of Sub-massive Pulmonary Embolism
Brief Title: ULTrasound Accelerated ThrombolysIs of PulMonAry Embolism
Acronym: ULTIMA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Collaborators: EKOS Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EKOS Protocol Number 08
Record Dates: First submitted 2010-07-15; First posted 2010-07-21 (Estimated); Results first posted 2016-10-18 (Estimated); Last update posted 2021-07-19 (Actual); Status verified 2021-07

CONDITIONS: Submassive Pulmonary Embolism
Keywords: Pulmonary embolism; Pulmonary thromboembolism; anticoagulation; thrombolysis; ultrasound accelerated thrombolysis
MeSH Terms: conditions — Pulmonary Embolism | interventions — Heparin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ultrasound accelerated thrombolysis (Experimental): Patients in this arm will receive anti-coagulation (intravenous unfractionated heparin) plus the EkoSonic Endovascular System will be used to deliver a low dose <20mg rt-PA (Actilyse) directly into the occlusive pulmonary thrombus.
  Interventions: Device: EkoSonic Endovascular System
- Intravenous unfractionated heparin (Active Comparator): Patients in this arm will receive the standard of care: intravenous unfractionated heparin used as anti-coagulation treatment.
  Interventions: Drug: Unfractionated heparin

INTERVENTIONS:
Device: EkoSonic Endovascular System — The EkoSonic Endovascular System will be used to deliver < 20 mg of rt-PA ( Actilyse) directly into the occlusive pulmonary thrombus.
  Arms: Ultrasound accelerated thrombolysis
Drug: Unfractionated heparin — Intravenous unfractionated heparin used for anticoagulation treatment
  Arms: Intravenous unfractionated heparin

SUMMARY:
The ULTIMA study is intended to prove that in patients with pulmonary embolism and a right ventricular end diastolic diameter to left ventricular end diastolic diameter ratio ≥1 (RV/LV ratio) will benefit from treatment with ultrasound accelerated thrombolysis (rt-PA) as compared to unfractionated heparin anticoagulation. Specifically, at 24 hours the RV/LV ratio will be significantly reduced in the treatment arm compared to the control arm.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute PE symptoms < 14 days.
* Filling defect by contrast-enhanced chest CT in at least one main or proximal lower lobe pulmonary artery
* Right ventricular dysfunction confirmed by echocardiography where the RV/LV end diastolic diameter ratio is ≥ 1.0.

Exclusion Criteria:

* Age less than 18 years or greater than 80 years
* Index PE symptom duration > 14 days
* Insufficient echocardiographic image quality in the apical or subcostal four-chamber view that prohibits the measurement of the right and left ventricular end-diastolic dimensions
* Known significant bleeding risk
* Administration of thrombolytic agents, e.g., tissue plasminogen activator, streptokinase, or urokinase, within the previous 4 days
* Active bleeding
* Known bleeding diathesis
* Known coagulation disorder, platelet count < 100 000/mm3, or previous use of vitamin K antagonists with INR > 2.5
* History of any intracranial or intraspinal surgery or trauma or intracranial/intraspinal bleed
* Intracranial neoplasm, arteriovenous malformation, or aneurysm
* Recent (< 3 months) GI bleeding.
* Recent (< 3 months) internal eye surgery or hemorrhagic retinopathy; recent (< 10 days) major surgery, cataract surgery, trauma, CPR, obstetrical delivery, or other invasive procedure.
* Allergy, hypersensitivity, or thrombocytopenia from heparin, rt-PA, or iodinated contrast, except for mild-moderate contrast allergies for which steroid pre-medication can be used.
* Estimated glomerular filtration rate (eGFR) < 50 ml/min as calculated by the Cockroft formula.
* Hemodynamic collapse at presentation defined as: need for cardiopulmonary resuscitation; or systolic blood pressure < 90 mm Hg for at least 15 min, or drop of systolic blood pressure by at least 40 mm Hg for at least 15 min with signs of end organ hypoperfusion (cold extremities or low urinary output < 30 mL/h or mental confusion); or need for catecholamine administration to maintain adequate organ perfusion and a systolic blood pressure of > 90 mm Hg.
* Severe hypertension on repeated readings (systolic > 180 mmHg or diastolic > 105 mmHg).
* Pregnant, lactation or parturition within the previous 30 days (positive pregnancy test, women of childbearing age must be tested).
* Participating in any other investigational drug or device study.
* Life expectancy < 90 days.
* Inability to comply with study assessments (e.g. due to geographic distance).
* Previous enrollment in this study
* Any other condition that the investigator feels would place the patient at increased risk if the investigational therapy is initiated.
* Known right-to-left shunt, for example from large patent foramen ovale or atrial septal defect
* Large (>10 mm) right atrial or right ventricular thrombus

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2010-07; Primary Completion 2013-04 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nils Kucher, Prof Dr med, Principal Investigator — Inselspital Bern, Kliniken für Angiologie und Kardiologie
Locations (10):
- Germany (9):
  - Klinikum Lippe-Detmold, Detmold
  - Klinikum Dortmund gGmbH, Dortmund
  - Universitätsklinikum Carl Gustav Carus an der TU Dresden, Dresden
  - Universitätsklinikum der Ernst-Moritz-Arndt-Universität,, Greifswald
  - Universitätsklinikum Heidelberg, Heidelberg
  - Klinikum der Ludwig-Maximilians-Universität (LMU), München
  - Christliches Krankenhaus Quakenbrueck, Quakenbrück
  - Helios Klinikum Siegburg, Siegburg
  - SRH Zentralklinikum Suhl, Suhl
- Inselspital Bern, Kliniken fur Kardiologie and Angiologie, Bern, Switzerland

REFERENCES:
- [Derived] Kucher N, Boekstegers P, Muller OJ, Kupatt C, Beyer-Westendorf J, Heitzer T, Tebbe U, Horstkotte J, Muller R, Blessing E, Greif M, Lange P, Hoffmann RT, Werth S, Barmeyer A, Hartel D, Grunwald H, Empen K, Baumgartner I. Randomized, controlled trial of ultrasound-assisted catheter-directed thrombolysis for acute intermediate-risk pulmonary embolism. Circulation. 2014 Jan 28;129(4):479-86. doi: 10.1161/CIRCULATIONAHA.113.005544. Epub 2013 Nov 13. PMID 24226805

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Multi-center, Phase III study at 8 tertiary care hospitals in Germany and Switzerland
Pre-assignment Details: Acute symptomatic PE confirmed by contrast-enhanced computed tomography (CT) with embolus located in at least 1 main or proximal lower lobe pulmonary artery RV to left ventricular dimension (RV/LV) ratio ≥1 obtained from the echocardiographic apical 4-chamber view
Groups:
- Unfractionated Heparin (UFH) Alone: Patients in this arm received the standard of care: intravenous unfractionated heparin used as anticoagulation treatment.
- Unfractionated Heparin (UFH) + EkoSonic Procedure: Patients in this arm received anticoagulation (intravenous unfractionated heparin) plus the EkoSonic Endovascular System was used to deliver a low dose of <20mg rt-PA (Actilyse) directly into the occlusive pulmonary thrombus.
Period: Overall Study
Arm/Group | Unfractionated Heparin (UFH) Alone | Unfractionated Heparin (UFH) + EkoSonic Procedure
Started | 29 | 30
Completed | 27 | 30
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- UFH (Alone): Patients in this arm received the standard of care: intravenous unfractionated heparin used as anticoagulation treatment.
- UFH + EkoSonic Procedure: Patients in this arm received anticoagulation (intravenous unfractionated heparin) plus the EkoSonic Endovascular System was used to deliver a low dose of <20mg rt-PA (Actilyse) directly into the occlusive pulmonary thrombus.
- Total: Total of all reporting groups
Arm/Group | UFH (Alone) | UFH + EkoSonic Procedure | Total
Number analyzed (Participants) | 29 | 30 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.0 (13.4) | 64.1 (15.2) | 63.1 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 19 | 31
  Male | 17 | 11 | 28

OUTCOME MEASURES:

1. Primary Outcome: Reduction of RV/LV Ratio
Description: Change in the end-diastolic RV/LV ratio from baseline to 24 hours by echocardiography.
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: Ratio
Groups:
- Unfractionated Heprin + EkoSonic Procedure: Patients in this arm received anti-coagulation (intravenous unfractionated heparin) plus the EkoSonic Endovascular System was used to deliver a low dose of <20mg rt-PA (Actilyse) directly into the occlusive pulmonary thrombus.
Arm/Group | Unfractionated Heparin (UFH) Alone | Unfractionated Heprin + EkoSonic Procedure
Number analyzed (Participants) | 28 | 25
Ratio | 0.03 (0.16) | 0.30 (0.20)

2. Primary Outcome: Major Bleeding and Intracranial Bleeding at 30 Days.
Description: Bleeding will be classified as major if it is associated with a fall in the hemoglobin level of at least 2.0 g/dl, transfusion of ≥ 2 units of red blood cells, or involvement of a critical site (e.g., intracranial, intraspinal). To aid in evaluating the relationship of bleeding events to rt-PA administration, they will also be categorized by whether they occurred within 3 days after the initiation of thrombolytic therapy.
Time Frame: 30 days
Measure: Number; unit: participants
Arm/Group | Ultrasound Accelerated Thrombolysis | Intravenous Unfractionated Heparin
Number analyzed (Participants) | 29 | 30
participants | 0 | 0

ADVERSE EVENTS:
Groups:
- UFH + EkoSonic: Patients in this arm received anticoagulation (intravenous unfractionated heparin) plus the EkoSonic Endovascular System was used to deliver a low dose of <20mg rt-PA (Actilyse) directly into the occlusive pulmonary thrombus.
Arm/Group | Unfractionated Heparin (UFH) Alone | UFH + EkoSonic
Serious Adverse Events (participants affected / at risk) | 4/29 | 3/30
Other Adverse Events (participants affected / at risk) | 2/29 | 0/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Unfractionated Heparin (UFH) Alone (N=29) | UFH + EkoSonic (N=30)
Postoperative wound infection (Surgical and medical procedures) | 0 | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Radius fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Supraventricular tachycardia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Bronchopneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Unfractionated Heparin (UFH) Alone (N=29) | UFH + EkoSonic (N=30)
Oedema peripheral (General disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days